CLINICAL TRIAL: NCT03227406
Title: The Evolution of Memories Across Wake and Sleep
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Beth Israel Deaconess Medical Center (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Robert Stickgold, Professor of Psychiatry, Beth Israel Deaconess Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 2016P000222; R01MH048832 (NIH)
Record Dates: First submitted 2017-07-19; First posted 2017-07-24 (Actual); Last update posted 2023-02-03 (Actual); Status verified 2023-02

CONDITIONS: Sleep Deprivation; Sleep
Keywords: sleep; memory; REM sleep; slow wave sleep; cognition; sleep spindles
MeSH Terms: conditions — Sleep Deprivation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Daytime Wake (No Intervention): Subjects are trained and retested during a single period of daytime wake
- Overnight sleep (No Intervention): Subjects are trained on one day and tested the next day, after a night of normal sleep
- Sleep deprivation (Experimental): Subjects are trained on one day and tested the next day, after a night of sleep deprivation
  Interventions: Behavioral: Sleep deprivation
- Daytime Nap (Experimental): Subjects are trained and then retested after a daytime nap
  Interventions: Behavioral: Nap

INTERVENTIONS:
Behavioral: Sleep deprivation — Subjects are kept awake all night.
  Arms: Sleep deprivation
Behavioral: Nap — Participants are given a 90-minute nap opportunity in the early afternoon.
  Arms: Daytime Nap

SUMMARY:
To further understanding of the relationship between sleep and memory the investigators will address and attempt to answer three questions, (1) how memories evolve across wake and sleep, (2) how different aspects of this memory evolution are reflected both behaviorally and in the EEG signal, and (3) what stages and features of sleep affect memory evolution. Together, these studies will provide a greater breadth and depth of knowledge concerning sleep's role in memory consolidation. Such knowledge would be of practical importance for educational practices, whether in schools, on the job, or in the military, and would also provide valuable information to the fields of sleep medicine and psychiatry, where interactions between sleep disorders and cognitive functioning are of great importance.

DETAILED DESCRIPTION:
Goal 1: How do memories evolve across wake and sleep? The investigators are interested in how specific memories are selected for change across periods of wake and sleep, and in characterizing the manner in which those memories change. There has been research into broad areas of memory, such as procedural and declarative memory, but other forms of memory, such as semantic memory, remain unexplored, as well as different subtypes of memory within these broad areas. Additionally, it is presently unknown how memories are selected for subsequent processing during sleep and wake. The investigators aim to characterize which memories change, how they are selected, and how they change differently over periods that include sleep versus periods during which participants remain awake.

Goal 2: How are these changes reflected behaviorally and in the EEG signal? The investigators will employ and develop specific behavioral and electrophysiological tasks and measures that allow one to probe the state of a particular type of memory and determine how it changes over periods of wake and sleep. EEG signals may be informative about the status of a memory during behavioral performance as well as during both waking and sleeping offline states.

Goal 3: What stages and features of sleep affect memory evolution? In the cases in which sleep in particular is found or suspected to influence memories in a unique way, the investigators will assess which stages and features of sleep are involved in that evolution. Generally, this will be accomplished by correlating measures such as time spent in a sleep stage, prominence of particular brain oscillations, or density of spindles with changes in behavior or in other EEG metrics

ELIGIBILITY:
Inclusion Criteria:

* willing and able to follow the protocol
* willing to refrain from alcohol and recreational drugs for the duration of the protocol
* in some cases, English as a first language, normal hearing, and/or normal or corrected to normal vision is required

Exclusion Criteria:

* self-reported sleep disturbances
* a history of mental illness
* the use of any drugs that could affect either sleep or cognitive functioning (e.g., sleeping pills or antidepressants)

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 276 (Actual)
Dates: Start 2016-03-01 (Actual); Primary Completion 2023-01-31 (Actual); Study Completion 2023-01-31 (Actual)

PRIMARY OUTCOMES:
Motor sequence task improvement | 4-24 hrs
  The increase in the number of correct sequences typed, from the last three training trials to the first three delayed-test trials, is calculated as a percent improvement.
Psychomotor vigilance task lapse rate | 4-24 hrs
  The absolute number of trials in a 5-min test period on which the participant fails to responds with 500ms is calculated as the lapse rate.
Serial reaction time test improvement | 4-24 hrs
  At two time points, separated by a period of wake or sleep, the average reaction time to stimuli in repeated sequence blocks is subtracted from the average reaction time in random blocks. The percent increase in this difference, from the final blocks in the first test to the first blocks in the second test, is calculated as a percent improvement.
Visual discrimination task improvement | 4-24 hrs
  At two time points, separated by a period of wake or sleep, the interpolated stimulus-mask ISI corresponding to 80% accuracy on the texture discrimination task is determined, and task improvement is calculated as the difference between these thresholds, in ms.

SECONDARY OUTCOMES:
Sleep architecture (absolute times) | 4-24 hrs
  Sleep is recorded with standard polysomnography and the amount of time spent in each wake and sleep stage calculated.
Sleep architecture (percent times) | 4-24 hrs
  The percent of total sleep time spent in each sleep stage is calculated.
Spindle | 4-24 hrs
  The density of sleep spindles per minute of N2 sleep is calculated.
Sleep microstructure | 4-24 hrs
  The EEG spectral power is calculated for N2 and N3 sleep.

CONTACTS AND LOCATIONS:
Overall Officials: Robert Stickgold, PhD, Principal Investigator — Beth Israel Deaconess Medical Center
Locations (1):
- Robert Stickgold, Boston, Massachusetts, United States